CLINICAL TRIAL: NCT01655355
Title: Revision of the Hip Joint - Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: rivk-001-HMO-CTIL
Record Dates: First submitted 2012-07-30; First posted 2012-08-01 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Revision of the Hip Joint

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Revison of the hip joint

SUMMARY:
Between the years 1999-2011 70 patients went through a revision of the hip joint(revision after not successful Total or Partial Hip Replacement). During the revision the Acetabular implant was found to be stable and it was decided not to replace it. The polyethylene insert was replaced and was fixated using a cement. Our purpose is to evaluate the physical condition of these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients that underwent a revision of the hip replacement without removing the acetabular implant
2. Insert polyethylene with cement

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that underwent a revision of the hip replacement without removing the acetabular implant.
Sampling Method: Non-Probability Sample

PRIMARY OUTCOMES:
Quality of life
  Quality of life as measured by the SF12 questionnaire.

SECONDARY OUTCOMES:
Function
  Function as measured by the Haris Hip Score

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel